CLINICAL TRIAL: NCT07063953
Title: Effects of Egoscue Exercises on Pain, Range of Motion and Physical Function in Patients With Knee Osteoarthritis
Brief Title: Effects of Egoscue Exercises in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0146 Momina
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: Pain; Physical Function; Range of motion
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egoscue Exercises (Experimental): Warm Up Exercises (5 min) which includes Stretching ,Walking (Forward, Backward, Sideways), Arm Circles, Side bends, March on the spot, Knee lifts, Standing Gluteal Contractions , Sitting heel raises, Isolated hip flexor lifts on a towel, Supine groin stretch on towels, Static back, Sitting Knee Pillow Squeezes, Sitting floor, Progressive supine groin, Supine calf-hamstring stretch with a strap,Foot circles and point flexes, Cool Down and Breathing Exercises
  Interventions: Other: Egoscue Exercises
- Standard Physical Therapy (Active Comparator): Hot pack & Transcutaneous Electric Nerve Stimulation (TENS) Myofascial Release Mulligan Mobilization with Movement Exercises
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Other: Standard Physical Therapy — Hot pack & Transcutaneous Electric Nerve Stimulation (TENS) Myofascial Release Mulligan Mobilization with Movement Exercises
  Arms: Standard Physical Therapy
Other: Egoscue Exercises — Warm Up Exercises (5 min) which includes Stretching ,Walking (Forward, Backward, Sideways), Arm Circles, Side bends, March on the spot, Knee lifts, Standing Gluteal Contractions , Sitting heel raises, Isolated hip flexor lifts on a towel, Supine groin stretch on towels, Static back, Sitting Knee Pillow Squeezes, Sitting floor, Progressive supine groin, Supine calf-hamstring stretch with a strap,Foot circles and point flexes, Cool Down and Breathing Exercises
  Arms: Egoscue Exercises

SUMMARY:
Knee osteoarthritis (KOA) is a chronic, debilitating illness with multiple etiologies that affects the entire knee joint. It is a leading cause of disability among the elderly population and necessitates effective interventions beyond pharmacotherapy due to the associated risks.

This study will address the existing literature gap by focusing on a novel therapeutic approach known as 'Egoscue Exercises', for managing knee osteoarthritis in the affected population.

DETAILED DESCRIPTION:
This Randomized Controlled Trial will be conducted at Riphah Rehab Training and Research Center, Lahore and District Health Quarter Hospital (DHQ), Sahiwal in a time span of 8 months. A sample of 42 participants aged 45-65 years, diagnosed with Grade 02 and 03 Knee Osteoarthritis, will undergo a comprehensive physiotherapy protocol, which includes standard physiotherapy knee OA treatment, either alone or in combination with Egoscue exercises. Participants will receive a minimum of 3 sessions per week, across four weeks.

Randomization, conducted by computer-generated stratified randomization, will ensure unbiased allocation to the two groups. Data collection will be carried out at baseline, 2 weeks, and 4 weeks, and includes outcomes in the form of pain measured by Numeric Pain Rating Scale (NPRS), range of motion measured by Goniometer, and physical function evaluated by Western Ontario and McMaster Universities Arthritis (WOMAC) index. The single-blind study will incorporate rigorous statistical analysis, using IBM SPSS software, version 25 for descriptive statistics, normality, and intergroup differences via t-tests and U tests.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 45 and 65 years ,
* Both genders male and female ,
* BMI ˃ 25 , and Knee OA clinically or radiologically diagnosed by Kellgren-Lawrence Method, Grade II and III

Exclusion Criteria:

* Age less than 45 years or older than 65 years,
* BMI < 25, Knee OA in grade I and IV, and
* Patients on steroid therapy and intra articular injection

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | upto 4 weeks
  The range of motion will be measured by using Universal Goniometer, which is a highly reliable and valid tool. It will measure knee joint range of motion which includes knee flexion and extension.
Western Ontario and McMaster Universities Arthritis (WOMAC) index | upto 4 weeks
  WOMAC Index is widely used in the evaluation of Knee Osteoarthritis. It is a 24 item questionnaire divided into 3 subscales:
  1. Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  2. Stiffness (2 items): after first waking and later in the day
  3. Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  The Numeric Pain Rating Scale (NPRS) is perhaps the most frequently applied scale used to quantify pain intensity in the clinical setting. It is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Basharat Hospital, Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma L. Osteoarthritis of the Knee. N Engl J Med. 2021 Jan 7;384(1):51-59. doi: 10.1056/NEJMcp1903768. No abstract available. PMID 33406330
- [Background] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Background] Giorgino R, Albano D, Fusco S, Peretti GM, Mangiavini L, Messina C. Knee Osteoarthritis: Epidemiology, Pathogenesis, and Mesenchymal Stem Cells: What Else Is New? An Update. Int J Mol Sci. 2023 Mar 29;24(7):6405. doi: 10.3390/ijms24076405. PMID 37047377
- [Background] Kondal S, Kulkarni V, Gaikwad A, Kharat A, Pant A. Automatic Grading of Knee Osteoarthritis on the Kellgren-Lawrence Scale from Radiographs Using Convolutional Neural Networks [Internet]. arXiv.org. 2020 [cited 2024 Jun 25].
- [Background] Yunus MHM, Nordin A, Kamal H. Pathophysiological Perspective of Osteoarthritis. Medicina (Kaunas). 2020 Nov 16;56(11):614. doi: 10.3390/medicina56110614. PMID 33207632
- [Background] Siddiq MAB, Clegg D, Jansen TL, Rasker JJ. Emerging and New Treatment Options for Knee Osteoarthritis. Curr Rheumatol Rev. 2022;18(1):20-32. doi: 10.2174/1573397117666211116111738. PMID 34784876